CLINICAL TRIAL: NCT03376932
Title: A Randomised Open-label Study to Compare the Effectiveness of the Fixed Dose Combination of FF/UMEC/VI (Using the Connected Inhaler System) With the Combination of FP/SAL Plus Tiotropium (Without the Connected Inhaler System) in Participants With Inadequately Controlled Asthma
Brief Title: Effectiveness of Fluticasone Furoate/ Umeclidinium/ Vilanterol (FF/UMEC/VI) Using the Connected Inhaler System (CIS) as Compared With Fluticasone Proprionate/ Salmeterol (FP/SAL) Plus Tiotropium (TIO) in Inadequately Controlled Asthma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawn due to internal reasons
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206821; 2017-001532-19 (EudraCT Number)
Record Dates: First submitted 2017-12-01; First posted 2017-12-19 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: Vilanterol; Fluticasone furoate; Connected Inhaler System; Dry powder inhaler; Umeclidinium; Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; Albuterol; Metered Dose Inhalers

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to receive either FF/UMEC/VI via the ELLIPTA DPI with the CIS or FP/SAL via the DISKUS DPI plus TIO via the RESPIMAT inhaler.
Masking Description: This will be an open-label study. Hence, masking will not be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Subjects receiving FF/UMEC/VI (100/62.5/25) mcg+ CIS (Experimental): Eligible subjects will receive SITT of FF/UMEC/VI based on their pre-study ICS dosage strength (mid- or high-dose). Subjects receiving mid-dose of ICS during pre-study will be administered with FF/UMEC/VI (100/62.5/25) mcg inhalation powder via ELLIPTA DPI, once daily in the morning or evening with the CIS. Subjects will also receive albuterol/salbutamol metered dose inhalers (MDIs) as a rescue medication throughout the study.
  Interventions: Drug: FF/UMEC/VI; Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: Metered Dose Inhaler; Device: Connected Inhaler System
- Subjects receiving FF/UMEC/VI (200/62.5/25) mcg+ CIS (Experimental): Eligible subjects will receive SITT of FF/UMEC/VI based on their pre-study ICS dosage strength (mid- or high-dose). Subjects receiving high-dose of ICS during pre-study will be administered with FF/UMEC/VI (200/62.5/25) mcg inhalation powder via ELLIPTA DPI, once daily in the morning or evening with the CIS. Subjects will also receive albuterol/salbutamol MDI as a rescue medication throughout the study.
  Interventions: Drug: FF/UMEC/VI; Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: Metered Dose Inhaler; Device: Connected Inhaler System
- Subjects receiving FP/SAL(250/50) mcg + TIO 5 mcg (Active Comparator): Eligible subjects will receive MITT of FP/SAL+ TIO based on their pre-study ICS dosage strength (mid- or high-dose). Subjects receiving mid-dose of ICS during pre-study will be administered with FP/SAL (250/50) mcg inhalation powder via DISKUS DPI with sensor, twice daily in the morning or evening plus TIO 5 mcg via RESPIMAT inhaler without sensor, once daily in the morning or evening. Subjects will also receive albuterol/salbutamol MDI as a rescue medication throughout the study.
  Interventions: Drug: FP/SAL; Drug: Tiotropium; Drug: Albuterol/salbutamol; Device: DISKUS DPI; Device: RESPIMAT inhaler; Device: Metered Dose Inhaler
- Subjects receiving FP/SAL(500/50) mcg + TIO 5 mcg (Active Comparator): Eligible subjects will receive MITT of FP/SAL+ TIO based on their pre-study ICS dosage strength (mid- or high-dose). Subjects receiving high-dose of ICS during pre-study will be administered with FP/SAL (500/50) mcg inhalation powder via DISKUS DPI with sensor, twice daily given in the morning or evening plus TIO 5 mcg via RESPIMAT inhaler without sensor, once daily in the morning or evening. Subjects will also receive albuterol/salbutamol MDI as a rescue medication throughout the study.
  Interventions: Drug: FP/SAL; Drug: Tiotropium; Drug: Albuterol/salbutamol; Device: DISKUS DPI; Device: RESPIMAT inhaler; Device: Metered Dose Inhaler

INTERVENTIONS:
Drug: FF/UMEC/VI — FF/UMEC/VI will be given as dry white powder delivered via the ELLIPTA DPI once daily in the morning or evening. The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 100 mcg or 200 mcg in each blister and the second strip contains UMEC 62.5 mcg and VI 25 mcg in each blister.
  Arms: Subjects receiving FF/UMEC/VI (100/62.5/25) mcg+ CIS; Subjects receiving FF/UMEC/VI (200/62.5/25) mcg+ CIS
Drug: FP/SAL — FP/SAL will be given as dry white powder delivered via the DISKUS DPI twice daily in the morning or evening. The DISKUS DPI holds a single blister strip with 60 blisters, which contains FP 250 mcg or 500 mcg and SAL 50 mcg per blister.
  Arms: Subjects receiving FP/SAL(250/50) mcg + TIO 5 mcg; Subjects receiving FP/SAL(500/50) mcg + TIO 5 mcg
Drug: Tiotropium — TIO will be given as clear, colorless, inhalation solution delivered via RESPIMAT inhaler once daily in the morning or evening. The RESPIMAT inhaler will contain 60 puffs with 2.5 mcg TIO per puff.
  Arms: Subjects receiving FP/SAL(250/50) mcg + TIO 5 mcg; Subjects receiving FP/SAL(500/50) mcg + TIO 5 mcg
Drug: Albuterol/salbutamol — Albuterol/salbutamol will be delivered as a rescue medication via MDI.
Device: ELLIPTA DPI — The ELLIPTA device will be used to administer FF/UMEC/VI once daily. The ELLIPTA DPI is a molded plastic two-sided inhaler that can hold two individual blister strips, which contain powder formulation for oral inhalation.
  Arms: Subjects receiving FF/UMEC/VI (100/62.5/25) mcg+ CIS; Subjects receiving FF/UMEC/VI (200/62.5/25) mcg+ CIS
Device: DISKUS DPI — The DISKUS device will be used to administer FP/SAL twice daily. The DISKUS DPI is a plastic inhalation delivery system containing a single-foil blister strip of a powder formulation of FP/SAL for oral inhalation.
  Arms: Subjects receiving FP/SAL(250/50) mcg + TIO 5 mcg; Subjects receiving FP/SAL(500/50) mcg + TIO 5 mcg
Device: RESPIMAT inhaler — The RESPIMAT inhaler will be used to administer TIO once daily. The RESPIMAT inhaler has a solution filled into a polyethylene/polypropylene cartridge with a polypropylene cap with integrated silicone sealing ring. The cartridge is enclosed within an aluminum cylinder.
  Arms: Subjects receiving FP/SAL(250/50) mcg + TIO 5 mcg; Subjects receiving FP/SAL(500/50) mcg + TIO 5 mcg
Device: Metered Dose Inhaler — Albuterol/salbutamol will be delivered as a rescue medication via MDI.
Device: Connected Inhaler System — The CIS will consist of a sensor, which clips on to the ELLIPTA DPI. This will inform subject's if/when they have taken their medication that is in the ELLIPTA inhaler. The sensor will measure when the ELLIPTA inhaler mouth piece cover is fully opened and closed and this data can be fed back, via the app on a mobile device to the subject. The sensors, app, and provider portal that provide data are subsequently described as the CIS.
  Arms: Subjects receiving FF/UMEC/VI (100/62.5/25) mcg+ CIS; Subjects receiving FF/UMEC/VI (200/62.5/25) mcg+ CIS

SUMMARY:
Asthma is a common, chronic respiratory disease affecting 1-18 percent of the population. It is accepted that much of the uncontrolled asthma is due to poor adherence and asthma outcomes in such cases may improve simply by increasing adherence to available treatments. GlaxoSmithKline (GSK) has developed a sensor, which clips on to the ELLIPTA® dry powder inhaler (DPI). This will inform subjects if/when they have taken their medication that is in the ELLIPTA inhaler, as well as other information, including: asthma management strategies, tracking of symptoms, asthma triggers, medication reminders and daily asthma forecasts. The sensors, application (app), and provider portal that provide data are subsequently described as the CIS. The combination of once-daily FF/UMEC/VI with the CIS will improve the disease management and adherence. Thus, this study is designed to study the effectiveness and adherence of single inhaler triple therapy (SITT) of FF/UMEC/VI with the CIS as compared to multiple inhaler triple therapy (MITT) of the combination of FP/SAL plus TIO without CIS in subjects with inadequately controlled asthma. The study randomization will be stratified by pre-study inhaled corticosteroids (ICS) dosage strength (mid- or high-dose). Subjects will be randomized in a 1:1 ratio to receive either FF/UMEC/VI delivered via the ELLIPTA DPI with the CIS or FP/SAL delivered via the DISKUS® DPI (with sensor only) plus TIO delivered via the RESPIMAT inhaler (without sensor). The maximum study duration will be approximately 29 weeks, which comprised of prescreen/ screening/ randomization period of up to 4 weeks, 24-week treatment period and a 1-week follow-up period. Approximately 1006 subjects will be randomized in the study. ELLIPTA and DISKUS are registered trademarks of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have their own Android or iPhone operating system (IOS) mobile device (example given [e.g.] smart phone or tablet) and a data package suitable for the installation and running of the app and sending and receiving data. Data used by the CIS is approximately 1 megabyte (MB) per month as a maximum; this is less data than a 1 minute video streamed from YouTube (2MB).
* Subjects must be willing and able to download the app on their personal mobile device and keep it turned on for the duration of the study. This will also require Bluetooth to be turned on for duration of the study. Subjects will also have to turn on mobile data for the app for the duration of study; unless travelling and when extra data roaming costs could be incurred.
* Subjects must be 18 years of age or older at the time of signing the informed consent.
* Subjects with a documented diagnosis of asthma by a respiratory physician or subjects with a documented asthma diagnosis by their general practitioner (GP) are required to have spirometry consistent with the diagnosis of asthma (e.g., reduced FEV1, reduced FEV1/forced vital capacity (FVC), or variable airflow obstruction) at or before Visit 0.
* Subjects who are able to perform spirometry that conforms to American Thoracic Society/ European Respiratory Society(ATS/ERS) technical standards at Visit 0 or Visit 1.
* Subjects are eligible if they require daily ICS/ long-acting beta-agonist (LABA) therapy (with a stable total daily dose of ICS of >250 microgram per day [mcg/day] FP, or equivalent) for at least 4 weeks prior to screening. Dosing regimen (once or twice daily to equal the total daily dose) should be restricted to the current local product labels/treatment guidelines.
* Subjects with inadequately controlled asthma (ACT total score <20) despite ICS/LABA maintenance therapy at Visit 1.
* Male or Female subjects will be included in the study. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) or A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 5 days after the last dose of study treatment. The Investigator is responsible for ensuring that subject understands how to properly use these methods of contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Subjects with current evidence of pneumonia, active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases, or other active pulmonary diseases including chronic obstructive pulmonary disease (COPD) or abnormalities other than asthma.
* Subjects with historical or current evidence of uncontrolled or clinically significant disease. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation (e.g. very low body mass index [BMI] or severely malnourished), or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Subjects with any of the following at screening would be excluded: myocardial infarction or unstable angina in the last 6 months; unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure.
* Moderate or severe hepatic impairment in subjects receiving high dose ICS.
* Subjects with a history of allergy or hypersensitivity to any corticosteroid, anticholinergic/ muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate are excluded from participation in this study.
* Subjects with a medical condition such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction should only be included if in the opinion of the Investigator the benefit outweighs the risk and that the condition would not contraindicate study participation.
* Subjects with active uncontrolled psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* 30 days or within 5 drug half-lives of the investigational drug (whichever is longer).
* Subjects who are medically unable to withhold their albuterol/salbutamol for the 6-hour period required prior to spirometry testing at each study visit.
* Smokers will be excluded as follows: current smokers (defined as subjects who have used inhaled tobacco products within the 12 months prior to screening [that is {i.e.}, cigarettes, e-cigarettes/vaping, cigars or pipe tobacco]); former smokers with a smoking history of >=10 pack years (e.g., >=20 cigarettes/day for 10 years).
* Subjects unable to comply with the study procedures due to infirmity, disability, or geographic location.
* Study Investigators, sub-Investigators, study coordinators, employees of a participating Investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Subjects who have taken part in more than 1 clinical trial in the 12 months prior to Visit 1 and/or subjects who have taken part in any of the following clinical trials in the 12 months prior to Visit 1: a clinical trial including audio and/or visual reminders for the subject to take their study treatment; any clinical trial during the 4 weeks prior to Visit 1;GSK study 207040.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-18 (Estimated); Primary Completion 2021-02-03 (Estimated); Study Completion 2021-02-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who have an asthma control test (ACT) total score of >=20 | Up to 24 weeks
  The ACT is a self-administered tool to identify subjects with poorly controlled asthma. It is a 5-item questionnaire measuring the frequency of shortness of breath, general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall assessment of asthma control. The response options for all these questions consist of a 5-point scale, ranging from 1 (all the time or not controlled at all for symptoms/activities) to 5 (not at all or completely controlled).
Percentage of subjects with an increase from Baseline of >=3 in ACT total score | Baseline and up to 24 weeks
  The ACT is a self-administered tool to identify subjects with poorly controlled asthma. It is a 5-item questionnaire measuring the frequency of shortness of breath, general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall assessment of asthma control. The response options for all these questions consist of a 5-point scale, ranging from 1 (all the time or not controlled at all for symptoms/activities) to 5 (not at all or completely controlled).

SECONDARY OUTCOMES:
Annualized rate of moderate and/or severe asthma exacerbations | Up to 24 weeks
  Annualized rate of moderate/severe asthma exacerbations will be compared to evaluate the effectiveness of FF/UMEC/VI with CIS on improving asthma control compared with FP/SAL+TIO after 24 weeks of treatment. Moderate asthma exacerbation is defined as deterioration in asthma symptoms, deterioration in lung function, or increased rescue bronchodilator use lasting for at least 2 days or more. Severe asthma exacerbation is defined as the deterioration of asthma requiring the use of systemic corticosteroids, or an increase from a stable maintenance dose, for at least 3 days or an inpatient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
Percentage of subjects who have a decrease from Baseline of >=4 in St George's Respiratory Questionnaire (SGRQ) total score | Baseline and up to 24 weeks
  The SGRQ is designed to measure quality of life in subjects with diseases of airway obstruction, measuring symptoms, impact, and activity. It is a well-established instrument, comprising 50 questions to be self-completed by the subject. Higher scores indicate worse health status, and a change of 4 points is considered a clinically relevant change.
Percentage of ELLIPTA versus DISKUS doses taken as prescribed over the 24-week treatment period | Up to 24 weeks
  The number of ELLIPTA and DISKUS doses taken will be collected using clip on sensors attached to the inhalers. The sensors will record the precise time and date when the mouthpiece cover of the inhalers has been opened and closed. Adherence is defined as the percentage of ELLIPTA and DISKUS doses taken as prescribed over the study treatment period as determined by the maintenance sensor records of date and time (within a 24-hour time period/window).
Change from Baseline in trough forced expiratory volume in 1 second (FEV1) | Baseline and up to 24 weeks
  FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on treatment is defined as the mean FEV1 value obtained prior to the last dose of investigational product.
Number of subjects with serious adverse events (SAEs) including hospitalizations for asthma | Up to 29 weeks from screening
  Any untoward event resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as an SAE. Number of subjects with incidences and type of SAEs including hospitalizations for asthma will be evaluated.
Number of subjects with AEs leading to withdrawal or discontinuation of treatment | Up to 25 weeks
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Number of subjects with AEs leading to withdrawal or discontinuation of treatment will be evaluated.
Number of subjects with AEs leading to dose modification | Up to 25 weeks
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Number of subjects with AEs leading to dose modification will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162